CLINICAL TRIAL: NCT05201092
Title: Interventional, Open-Label, Single-Dose Study Investigating the Absorption, Metabolism and Excretion (AME) of Lu AG06466 Following Oral Dosing of 14C-Lu AG06466 to Healthy Men
Brief Title: A Study Investigating Lu AG06466 in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19960A; 2021-002048-54 (EudraCT Number)
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-Lu AG06466 (Experimental): Participants will receive a single oral dose of [14C]-Lu AG06466 on Day 1 in the fed state.
  Interventions: Drug: [14C]-Lu AG06466

INTERVENTIONS:
Drug: [14C]-Lu AG06466 — [14C]-Lu AG06466 will be administered per schedule specified in the arm description.

SUMMARY:
The purpose of this study is to investigate how the drug Lu AG06466 is absorbed, metabolized, and excreted from the body, for example, what the body does to the drug after swallowing a single dose.

DETAILED DESCRIPTION:
Researchers will measure the levels of the drug and its breakdown product in each participants blood for up to 5 days after dosing. Radioactivity in urine and feces will be measured for up to 3.5 weeks after dosing.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30 kilograms (kg)/square meter (m^2) and a body weight of ≥60 kg at the Screening Visit and at the Baseline Visit.
* The participant has a resting supine systolic blood pressure ≥91 and ≤140 millimeters of mercury (mmHg) and a resting supine diastolic blood pressure ≥51 and ≤85 mmHg at the Screening Visit and at the Baseline Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, neurological examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has taken disallowed medication <1 week prior to the first dose of study drug or <5 half-lives prior to the Screening Visit for any medication taken.
* The participant has orthostatic hypotension, defined as a decrease in systolic blood pressure ≥20 mmHg or a decrease in diastolic blood pressure ≥10 mmHg from supine to standing, at the Screening Visit or at the Baseline Visit.
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.
* The participant has received a COVID-19 vaccination less than 30 days prior to the first dose of study drug.
* The participant trains/exercises intensively, for example, for a marathon or triathlon, or at a competitive level.
* The participant is exposed to significant levels of ionizing radiation at work.
* The participant has undergone any clinical procedures involving significant exposure to radiation (excluding dental X-ray and common X-rays of the chest or extremities) <12 months prior to the Screening Visit.
* The participant has received radiolabelled material <12 months prior to the Screening Visit.

Note: Other inclusion and exclusion criteria may apply.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
Cumulative Percent Recovery of Radioactivity in Urine | From Day 1 to Day 23
Cumulative Percent Recovery of Radioactivity in Faeces | From Day 1 to Day 23
Total Cumulative Percent Recovery of Radioactivity in Urine and Faeces | From Day 1 to Day 23
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Lu AG06466 | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
AUC0-inf of Metabolite Lu AG06988 in Plasma | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Maximum Observed Concentration (Cmax) of Lu AG06466 in Plasma | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Cmax of Metabolite Lu AG0988 in Plasma | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Time to Reach Cmax (tmax) of Lu AG06466 | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Tmax of Metabolite Lu AG06988 | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Apparent Elimination Half-life (t1/2) of Lu AG06466 in Plasma | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
t1/2 of Metabolite Lu AG06988 in Plasma | 0 (predose) up to 96 hours postdose on Day 1 to Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- LabCorp Clinical Research Unit Ltd, Leeds, United Kingdom